CLINICAL TRIAL: NCT05757856
Title: An Open-label Phase 2 Study Assessing the Safety, Tolerability and Preliminary Diagnostic Performance of a Radioactive Imaging Agent, NDX-3315 and NDX-3324, in Healthy Adult Participants and Patients With Eosinophilic Esophagitis
Brief Title: A Study to Investigate Safety and Tolerability of NDX-3315 and NDX-3324 in Healthy Participants and Patients With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NexEos Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NDX-3315-1001
Record Dates: First submitted 2023-02-10; First posted 2023-03-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; EoE; Diagnostic
MeSH Terms: conditions — Eosinophilic Esophagitis; Disease

STUDY DESIGN:
Intervention Model Description: Open-label single-arm study.
Masking Description: The pathologist and immunostaining analyst receiving study participant biopsies for analysis, as well as the radiologist scoring the scans will be blinded to EoE diagnosis and other test results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regimen 10 (Reclined) (Experimental): NDX-3315 or NDX-3324 delivered via oral syringe at ~ 1.5 mL per minute while sitting reclined.
  Interventions: Drug: NDX-3315 and NDX-3324

INTERVENTIONS:
Drug: NDX-3315 and NDX-3324 — Oral solution

SUMMARY:
An open-label phase 2 study to assess the safety and exploratory diagnostic performance of the oral radiopharmaceutical agent NDX-3315 and NDX-3324 in healthy participants and patients with eosinophilic esophagitis (EoE).

DETAILED DESCRIPTION:
This study is a multi-site, Phase 2, open-label study of orally administered NDX-3315 or NDX-3324 and esophageal imaging in healthy participants and participants with EoE.

Study details include:

* The study duration or period will be up to around 10 weeks.
* Participants will receive either one or two doses of NDX-3315 or NDX-3324 depending on their assigned regimen arm. EoE participants will receive two doses; healthy participants will receive one dose. There will be a SPECT/CT scan performed at each dose.
* The visit frequency will be three site visits for healthy participants and four site visits for EoE participants followed by one follow-up phone call visit within the study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants:

  • Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG) assessment.
* EoE Participants:

  * Documented diagnosis of EoE (based on prior endoscopy with biopsies showing eosinophils ≥15 / HPF); AND
  * History (by patient report) of recurrent dysphagia and/or other related EoE symptoms (with intake of solids off anti-inflammatory therapy) prior to screening; dysphagia is defined as trouble swallowing solid food, or having solid food stuck, by patient report.

Exclusion Criteria:

* Medical Conditions:

  * Participant with presence of any other disease of the GI tract, including cancer, autoimmune esophageal disease, GERD which is symptomatic or uncontrolled, Barrett's esophagus, eosinophilic gastritis, enteritis, colitis, or proctitis; inflammatory bowel disease; or celiac disease. Known motility disorder of esophagus; achalasia or suspicion thereof.
  * Sleep apnea, if considered by the investigator a concern for the endoscopic procedure.
  * History of recurrent aspiration pneumonia.
  * History of bleeding disorders, liver cirrhosis or esophageal varices.
  * A current malignancy or previous history of cancer in remission for less than 5 years prior to Screening (participants will not be excluded if they had localized carcinoma of the skin that was resected for cure).
  * Participant with a Body Mass Index >40 m2/kg or inability to undergo a CT (or SPECT scan) due to weight limitations.
  * Participant is pregnant or nursing.
* Prior/Concomitant Therapy:

  * Participant who is on anticoagulation therapy that, in the investigator or Medical Monitor's opinion, cannot safely come off medication.
  * Use of chronic aspirin (with the exception of low-dose aspirin as long as the dose remains stable and not increased while on study), nonsteroidal agents, or anti-coagulants within 2 weeks prior to screening.
  * Use of systemic corticosteroids within 3 months or swallowed topical corticosteroids within 6 weeks prior to Screening visit.
  * Participant is being treated with systemic immunosuppression, carafate (sucralfate), or investigational agent of any kind within less than 3 months or 5 half-lives, whichever is longer, prior to Screening visit (this also includes investigational formulations of marketed products).
* Diagnostic Assessments:

  * Evidence of clinically significant abnormality in the hematological and biochemical assessments at Screening Visit, specifically: International Normalized Ratio (INR) >1.4; platelet count <80,000/μL and creatinine level >2 mg/dL.
  * ECG: QTcF ≥450 msec for males and QTcF ≥470 msec for females at the time of screening.
* Other Exclusion Criteria:

  * Any condition that would not permit adequate biopsies of the esophagus (e.g., esophageal varices, significant stricture precluding passage of a 9 mm endoscope, known allergy to sedative used for endoscopy).
  * Healthy Participants Only: A history or current diagnosis of allergic diseases (Should be discussed with Medical Monitor and PI to decide whether exclusionary), autoimmune disease, chronic rhinosinusitis or serum immunoglobulin E (IgE) level ≥100 kU/L. On any medications including NSAIDS and any over the counter (OTC) medications unless it is birth control or acne medications with the exception of Accutane, or if deemed acceptable to use by Medical Monitor and PI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
The proportion of all participants with AEs following administration of NDX-3315 and NDX-3324 | From start of study drug administration up to End of Study (EOS) ( Up to 3 Weeks)
  An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product and that does not necessarily have causal relationship with this treatment.
Peak eosinophil counts per high-power field (HPF) | Up to 10 days after last dose
  A blinded pathologist will perform peak eosinophil counts per high-power field (HPF) on biopsy specimens of the esophagus.
Absolute quantification of SPECT imaging | Up to 45 minutes after dose
  SPECT images will be analyzed for radioactive per region of interest(ROI) of the esophagus.
Determine Concordance of Outcomes | Up to 10 Days After Last Dose
  Determine concordance rate between
  1. eMBP1 immunostaining score on biopsy specimens (esophagus) and
  2. NDX-3315 and NDX-3324 absolute quantification of SPECT imaging of esophagus

SECONDARY OUTCOMES:
Partial Thromboplastin Time (PTT) as marker of pharmacodynamics (PD) | Baseline, 2 hours post-dose (Up to 1 Week)
  Blood samples will be collected to measure Partial Thromboplastin Time (PTT), which is a blood test that looks at how long it takes for blood to clot.
Radioactivity of blood collected from participants exposed to NDX-3315 and NDX-3324. | 2.5 hours post-dose (Up to 1 Week)
  Blood samples will be collected to measure radioactivity as counts per minute(cpm) and disintegrations per minute(dpm).
Visual ratings of SPECT images | Up to 45 minutes after dose
  A blinded central reviewer will review SPECT images for uptake of NDX-3315 or NDX-3324 per region of interest(ROI) of the esophagus using a 5-point scale (0= no uptake to 4 = uptake similar to bowel), with 4 being the worst result.
Deposition of eMBP1 | Up to 10 days after last dose
  A blinded immunostaining analyst will perform analysis of deposition of Eosinophil Major Basic Protein 1 (eMBP1) via immunostaining of biopsy specimens of the esophagus.
EoE Endoscopic Reference Score (EREFS) | Up to 10 days after last dose
  The EoE-EREFS (Edema, Rings, Furrows, Exudates, Strictures) scores are used to measure the endoscopically identified EoE esophageal mucosal characteristics. The evaluation includes stricture (if applicable); exudates (absent, mild, severe); furrows (absent, present); edema (absent, present); crepe paper esophagus (absent, present), and overall general appearance incorporating all endoscopically-identified EoE findings (e.g., fixed rings, strictures, whitish exudates, furrowing, edema, and crepe paper mucosa). The EoE -EREFS score being used in this study has a range from 0-11, with 11 being the worst result.
EoE Symptom Collection Questionnaire | Baseline (All participants), Day 1 (EoE participants only)
  A questionnaire will be used to collect study participant symptoms such as severity of EoE dysphasia as well as concerns about pain. Answers will have corresponding score ranging from 1-18, with 18 being the worst result.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern Univerisity, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No